CLINICAL TRIAL: NCT03288818
Title: IIS: Phase II Study of Low Dose Total Skin Electron Beam Treatment (TSEBT) Followed by Maintenance Valchlor for Patients With Mycosis Fungoides
Brief Title: Low Dose Total Skin Electron Beam Radiation Therapy and Mechlorethamine Hydrochloride Gel in Treating Patients With Mycosis Fungoides
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding discontinued
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16C.514; JT 8557 (Other: JeffTrial Number)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Amines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- low dose TSEBT, mechlorethamine hydrochloride gel (Experimental): Patients undergo low dose TSEBT for 2 weeks. After 30 days of observation, patients receive mechlorethamine hydrochloride gel topically daily at week 7 and then once weekly up to week 54.
  Interventions: Drug: Mechlorethamine Hydrochloride Gel; Procedure: Total Skin Electron Beam Radiation Therapy

INTERVENTIONS:
Drug: Mechlorethamine Hydrochloride Gel — Given topically
  Other Names: Valchlor
Procedure: Total Skin Electron Beam Radiation Therapy — Undergo low dose (TSEBT) Total Skin Electron Beam Therapy
  Other Names: TSEB radiation therapy

SUMMARY:
This phase II trial studies how well low dose total skin electron beam radiation therapy and mechlorethamine hydrochloride gel work in treating patients with mycosis fungoides. Total skin electron beam radiation therapy uses high energy x-rays directed at the entire surface of the body to kill cancer cells and shrink tumors. Mechlorethamine hydrochloride gel may help patients in remission of disease, reduction in disease staging, and enhanced quality of life. Giving total skin electron beam radiation therapy and mechlorethamine hydrochloride gel may work better in treating patients with mycosis fungoides.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the time to progression of patients treated with total skin electron beam therapy (TSEBT) followed by the year-long maintenance mechlorethamine hydrochloride gel (Valchlor) regimen.

SECONDARY OBJECTIVES:

I. To assess the response rate (complete response [CR] and partial response [PR]) of patients treated with total skin electron beam therapy (TSEBT) followed by the year-long maintenance Valchlor regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of diagnosis as evidenced by one or more clinical features consistent with mycosis fungoides cutaneous T-cell lymphoma
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with requirements of the study
* Skin biopsy specimen of representative lesion obtained at screening of study and deemed diagnostic of mycosis fungoides by principal investigator
* Mycosis fungoides patients that have stage T2-4 N0-1 M0B0 disease
* Availability of subject to be observed for up to 18 months post-screening evaluation
* Life expectancy greater than 6 months

Exclusion Criteria:

* Pregnant or breast-feeding females
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data
* Patients diagnosed with Sezary syndrome; Sezary syndrome is equivalent to mycosis fungoides that develops to stage IVA/B with B2 (high blood tumor burden) involvement, and as such requires a more aggressive treatment regimen than Valchlor or TSEBT
* Underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of the patient to undergo treatment
* Minimum 3 weeks since prior systematic treatment or phototherapy
* Exclusion of people that do not understand the risks, such as decisionally-impaired individuals, prisoners, and vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | Up to week 54
  Will be evaluated using the Kaplan-Meier estimator of the survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Joya Sahu, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/